CLINICAL TRIAL: NCT06610357
Title: Evaluation of Long-Term Effects of Selective Dorsal Rhizotomy Surgery on Function and Mobility in Children With Cerebral Palsy Using the International Classification of Functioning, Disability, and Health (ICF) Model
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Neslihan Yildizdagi, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: NYildizdagii
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Diplegic Cerebral Palsy; Muscle Tone Abnormalities
Keywords: Cerebral Palsy; ICF; Muscle Tone; Mobility; Long-Term effects; Selective Dorsal Rhizotomy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with diparetic serebral palsy: 42 diparetic children with cerebral palsy were included in the study. The Modified Ashworth Scale (MAS), the Children's Functional Independence Measure (WeeFIM)-Mobility section and the Gross Motor Function Measure-88 (GMFM-88) were applied before and after SDR surgery.
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — 42 diparetic children with cerebral palsy were included in the study. The Modified Ashworth Scale (MAS), the Children's Functional Independence Measure (WeeFIM)-Mobility section and the Gross Motor Function Measure-88 (GMFM-88) were applied before and after SDR surgery.

SUMMARY:
Cerebral Palsy (CP) is a neurodevelopmental disorder characterized by abnormalities in muscle tone, movement, and motor skills as a result of permanent, non-progressive damage to the developing brain before, during, or after birth (Tedla & Reddy, 2021). The worldwide prevalence of CP is 2-3 per 1000 live births (Paul et al., 2022). The most common type is spastic type CP with a prevalence rate of 70-80% (Christensen et al., 2014). Spastic type CP is divided into three groups: diparetic (38%), hemiparetic (39%) and quadriparetic (23%) (Novak et al., 2014). In diparetic CP (DCP); lower extremity involvement is more prominent than upper extremity involvement (Elbasan et al., 2017). Selective Dorsal Rhizotomy (SDR) is a surgical technique applied for spasticity management in children with spastic diparetic CP (Novak et al., 2014). The positive effect of SDR on function and mobility has been proven (Novak et al., 2020). Studies in the literature have revealed the long-term effects of SDR through surveys. Many problems are observed in individuals with CP. It is very important to evaluate the situation in detail in order to analyze it well. It is recommended to use the International Classification of Functioning, Disability and Health (ICF) model, which creates a framework to evaluate children with a diagnosis of DCP in a healthy way and develop effective treatment strategies (Riyahi et al., 2024). ICF enables the identification of situations related to human functionality and limitations and creates a framework (Çankaya & Seyhan, 2016). The aim of this study is to evaluate the late effects of SDR surgery on function and mobility in cases with DCP using the ICF model.

DETAILED DESCRIPTION:
It's an observational study. Purpose of the study: This study aims to assess the long-term impact of SDR surgery on function and mobility in children with CP using the ICF model.

The study included 42 diparetic CP cases. These cases were aged between 2-9 years, with a mean age of 4.7±1.7 years.

* How did the long-term the Modified Ashworth Scale (MAS) values after SDR change compared to before the operation?
* How did the long-term the Gross Motor Function Measure-88 (GMFM-88) values after SDR change compared to before the operation?
* How did the long-term the Children's Functional Independence Measure (WeeFIM)- Mobility scores after SDR change compared to before the operation?

The Modified Ashworth Scale (MAS), the Gross Motor Function Measure-88 (GMFM-88) and the Children's Functional Independence Measure (WeeFIM)-Mobility section were applied to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Their ages must be between 0-17,
* They must be diagnosed with diparetic CP,
* The participants and their parents want to participate in the study voluntarily
* The Gross Motor Function Classification System (GMFSS) level II-IV
* Having a sitting level between 4-8 according to the Level Sitting Scale (LSS)
* Actively continuing the Physiotherapy and Rehabilitation (PTR) program for at least 2 months in the post-operative period.

Exclusion Criteria:

* Having different types of CP such as dyskinetic, ataxic and mixed type
* Having spastic quadriparetic or hemiparetic type of CP
* Having any surgical history on the musculoskeletal system,
* Having Botulinum Toxin injection within the last 6 months.

Ages: 0 Days to 17 Years | Sex: All
Age Groups: Child
Study Population: 42 children with Diparetic Cerebral Palsy were included in the study.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The Modified Ashworth Scale (MAS) | baseline
  It is used to describe the muscle's resistance to passive movement, the ease with which the joint can be moved within the available range. It is a 6-point scale that measures the muscle's resistance to passive movement by passively moving the joint through its possible normal range of motion. Within the scope of the study, lower extremity muscles; hip flexors, hip adductors, hip internal rotators, knee flexors, knee extensors and ankle plantar flexors will be evaluated with MAS.
The Gross Motor Function Measure-88 (GMFM-88) | baseline
  It is an observational scale developed to evaluate the gross motor skills of children with CP and identify limitations. Gross motor function is evaluated in 5 sections: supine position and rolling over, sitting, crawling and kneeling, standing and walking-running and jumping. It consists of a total of 88 items. Each item is scored as 0, 1, 2, 3 or "not tested" and the total score and percentage (%) are calculated.
The Children's Functional Independence Measure (WeeFIM) | baseline
  It was developed to evaluate the functional independence levels of children with developmental disorders in daily living activities. The scale consists of 6 parts: self-care (6 items), sphincter control (2 items), transfers (3 items), movement (2 items), communication (2 items), social and cognitive status (3 items). There are a total of 18 items in the sections. All items in the sections are scored between 1-7. 1 point, complete dependence; 7 points indicate complete independence. A total of minimum 18 (fully dependent) points and a maximum of 126 (fully independent) points can be obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, AA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.